CLINICAL TRIAL: NCT05269082
Title: In Vitro Assessment of Hypersensitivity to TAK-880 Compared to Gammagard S/D in Blood From Patients at Increased Risk of Developing Hypersensitivity Reactions
Brief Title: A Study to Assess the Hypersensitivity to TAK-880 Compared to Gammagard S/D in Blood of Children, Teenagers and Adults
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-880-5001
Record Dates: First submitted 2022-03-04; First posted 2022-03-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Drug Hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Pediatric and adult participants who are on Gammagard S/D prescribed for any approved indication will be enrolled in this cohort and evaluated during the observation period (approximately 6 months).
  Interventions: Other: No intervention
- Cohort 2: Pediatric and adult participants who were previously treated with Gammagard S/D prescribed for any approved indication and are on another human immunoglobulin treatment will be enrolled in this cohort and evaluated during the observation period (approximately 6 months).
  Interventions: Other: No intervention
- Cohort 3: Pediatric and adult primary immunodeficiency (PID) participants with immunoglobin A (IgA) deficiency who have a serum IgA level of less than (<) 7 milligrams per deciliter (mg/dL) (0.07 grams/liter [g/L]) or below the detectable limit and have received other therapies (prophylactic antibiotics or immunoglobulin treatment other than Gammagard S/D) will be enrolled in this cohort and evaluated during the observation period (approximately 6 months).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The aim of this study is to find out whether TAK-880 creates hypersensitivity reactions compared to Gammagard S/D by testing blood taken from participants who have a higher risk of becoming hypersensitive to immunoglobulin products.

This study is about collecting data available in the participant's medical record. No study medicines will be provided to participants in this study. Each participant will fill out a study questionnaire during a routine doctor visit. Blood will be taken from participants who have a higher risk of developing hypersensitivity reactions to immunoglobulin products.

ELIGIBILITY:
Inclusion criteria:

* At least 2 years of age except PID participants with selective IgA deficiency (the lower age limit in this group of participants is 4 years of age).
* Participant has previously received at least one infusion of Gammagard S/D prescribed for any approved indication (PID, B-cell Chronic Lymphocytic Leukemia, Idiopathic Thrombocytopenic Purpura, Kawasaki Syndrome) OR PID participant with IgA deficiency (serum IgA level of < 7 mg/dL (0.07 g/L) or below the detectable limit in participants older than 4 years) and has received other therapies (prophylactic antibiotics or immunoglobulin treatment other than Gammagard S/D).
* Participant/legally authorized representative is willing to sign an informed consent form or assent form as applicable and is able to comply with the requirements of the protocol.

Exclusion criteria:

-There are no applicable exclusion criteria for this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult participants who are at increased risk of developing hypersensitivity reactions who have been prescribed immunoglobulin treatments according to the investigator's judgment will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with In Vitro Hypersensitivity to TAK-880 in Comparison to Gammagard S/D | Up to approximately 6 months
  Levels of in vitro hypersensitivity to TAK-880 in comparison to a reference product (Gammagard S/D) using hypersensitivity assays to address (but not limited to) immune cell activation and cytokine secretion, stratified by anti-IgA antibody levels will be evaluated during the study. Number of participants with In vitro hypersensitivity to TAK-880 in comparison to Gammagard S/D will be reported.
Number of Participants with Drug Hypersensitive Reactions to Immunoglobulin Products for Cohort 1 and 2 | Up to approximately 6 months
  Number of Participants with drug hypersensitive reactions to immunoglobulin products who have previously received at least one infusion of Gammagard S/D in Cohorts 1 and 2 will be reported.
Number of Participants with History to Drug Hypersensitive Reactions | Up to approximately 6 months
  Number of participants with history to drug hypersensitive reactions will be reported.
Number of Participants Categorized by Clinical Characteristics | Up to approximately 6 months
  Number of participants categorized by clinical characteristics such as geographic location of residency, level of education will be reported.
Number of Participants Categorized by Treatment Patterns | Up to approximately 6 months
  Number of participants categorized by treatment patterns will be reported.
Health Related Quality of Life Measured by 36-Item Short Form Health Survey (SF-36) | Up to approximately 6 months
  SF-36 is a generic quality-of-life instrument that has been widely used to assess health-related quality of life (HRQL). SF-36 consists of 36 items that are aggregated into 8 multi-item scales (physical functioning [ranges from 1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]). Four domains comprised physical component summary (PCS) score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised mental component summary (MCS) score (vitality, social functioning, role-emotional, mental health). The total scores range from 0 to 100. Higher scores indicate better quality of life.
Health Related Quality of Life Measured by EuroQol 5 Dimensions Questionnaire (EQ-5D) | Up to approximately 6 months
  EQ-5D is a well-validated, general preference-based, health-related QoL instrument. The EQ-5D encompasses 5 domains, asking participants to rate their perceived health state today on the following dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each domain has 5 possible levels: "no problems" (Level 1), "slight problems" (Level 2), "moderate problems" (Level 3), "severe problems" (Level 4), and "extreme problems" (Level 5). Each domain is assigned a level, and levels are combined to create a 5-digit number describing the patient's health state. For each participant, an index value is determined from a published country-specific value set. This index value or utility score ranges from 0 to 1.00 (with 1.0 representing perfect health) and is used in the calculation of quality-adjusted life years (QALYs) that are used to inform economic valuations of health interventions. A positive change from baseline indicates improvement.
Health Related Quality of Life Measured by Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) Validated Instrument for Cohort 1 and 2 | Up to approximately 6 months
  TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness (3 items), convenience (3 items), and global satisfaction (3 items). Scores for each domain are calculated by adding up the items in each domain and then transforming the composite score into a value ranging from 0 to 100. Higher score indicated greater satisfaction in that domain.
Patient Reported Outcomes (PROs) Using PID-Specific Life Quality Index (LQI) Questionnaire for Cohort 1 and 2 | Up to approximately 6 months
  The PID-LQI questionnaire involves 15-items, divided into four domains: treatment interferences (6 items), therapy-related problems (4 items), therapy setting (3 items), and treatment costs (2 items). Items are rated on a 7-point Likert-type scale ranging from 1: "Extremely poor" to 7: "Extremely good". The items measure the impact of the treatment on patient quality of life: factor I (treatment interference), factor II (therapy-related problems), factor III (therapy settings). Results range from 0 (maximal concern) to 100 (no concern). PROs using PID-specific LQI questionnaire in Cohort 1 and 2 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- PPD, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/ad94e8b04ffb466a?idFilter=%5B%22TAK-880-5001%22%5D